CLINICAL TRIAL: NCT00119379
Title: Reversibility of Mitochondrial Toxicity in HIV Lipoatrophy
Brief Title: Effectiveness of Nucleoside Supplementation or Switch to Tenofovir in Reversing Fat Loss in HIV Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Grace McComsey, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI060484-01A2B; R01AI060484 (NIH)
Record Dates: First submitted 2005-07-11; First posted 2005-07-13 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections; Lipodystrophy; Metabolic Diseases; Nutrition Disorders
Keywords: lipoatrophy; mitochondria; HIV; treatment experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Metabolic Diseases; Nutrition Disorders | interventions — Uridine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- uridine supplementation (Experimental): NucleomaxX 36 grams TID every other day
  Interventions: Drug: NucleomaxX
- Switch to Tenofovir (Active Comparator): Switch of AZT or d4T to Tenofovir Disoproxil Fumarate
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: NucleomaxX — NucleomaxX 36 grams TID every other day
  Other Names: uridine
  Arms: uridine supplementation
Drug: Tenofovir Disoproxil Fumarate — Switch of thymidine nucleoside reverse transcriptase inhibitors to Tenofovir Disoproxil Fumarate
  Other Names: TDF
  Arms: Switch to Tenofovir

SUMMARY:
HIV lipoatrophy is a condition marked by fat loss; it occurs in many patients taking antiretroviral (ARV) therapy that includes nucleoside reverse transcriptase inhibitors (NRTIs). Lipoatrophy may be related to mitochondrial toxicity, a condition that can damage the heart, nerves, muscles, kidneys, and liver, and can affect the body's ability to produce energy. NucleomaxX is a food supplement consisting of a sugar cane extract high in nucleosides, which are building blocks that may counteract the negative effects of NRTIs. Tenofovir disoproxil fumarate (TDF) is an NRTI that may cause less lipoatrophy than other drugs in its class, such as zidovudine (ZDV) or stavudine (d4T). The purpose of this study is to determine whether nucleoside supplementation with NucleomaxX and substitution of TDF for ZDV or d4T in an ARV regimen can reverse fat loss caused by mitochondrial toxicity in HIV infected adults.

Study hypotheses: 1) The substitution of TDF for d4T or ZDV in patients with HIV lipoatrophy will result in an increase in mitochondrial DNA content in fat, skeletal muscle, and peripheral blood mononuclear cells (PBMCs), which in turn will lead to an improvement in mitochondrial function as assessed by electron transport chain (ETC) and oxidative phosphorylation pathway (OXPHOS) activity. The latter should lead to a decrease in fat apoptosis and in mitochondrial and lipid oxidative damage biomarkers. 2) Supplementation with uridine (via NucleomaxX) will increase mtDNA content in adipose tissue and increase body fat content.

DETAILED DESCRIPTION:
NRTIs are an important part of many ARV regimens used to treat HIV infected patients; however, the relationship between NRTI-induced mitochondrial dysfunction and lipoatrophy is still unclear and requires additional research. Additionally, the relationship between the gain in dual-energy x-ray absorptiometry (DEXA)-measured limb fat and mitochondrial DNA (mtDNA) content, mitochondrial function, fat apoptosis, and oxidative damage will also be examined in this study.

Patients will participate in this study for 48 weeks. Participants will be randomly assigned to one of two groups. Group 1 patients will receive NucleomaxX every other day. Group 2 patients will substitute TDF for ZDV or d4T every day in their current stable NRTI-containing ARV regimen. NucleomaxX will be provided to Group 1 patients, but TDF or any other ARV will not be provided by this study.

There will be 10 study visits, which will occur at study entry and Weeks 2, 4, 8, 12, 18, 24, 30, 36, and 48. Blood collection will occur at all visits. Additionally, urine collection, DEXA scans, and fat biopsies will be done at study entry and Weeks 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV lipoatrophy
* Receiving a stable stavudine- or zidovudine-containing ARV regimen
* HIV-1 RNA viral load less than 50 copies/ml

Exclusion Criteria:

* Coagulopathies or other bleeding disorders
* Diabetes requiring medication
* Creatinine clearance less than 50 ml/min
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace A. McComsey, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McComsey GA, O'Riordan M, Setzer B, Lebrecht D, Baron E, Walker UA. Uridine supplementation in HIV lipoatrophy: pilot trial on safety and effect on mitochondrial indices. Eur J Clin Nutr. 2008 Aug;62(8):1031-7. doi: 10.1038/sj.ejcn.1602793. Epub 2007 May 30. PMID 17538545
- [Derived] McComsey GA, O'Riordan M, Choi J, Libutti D, Rowe D, Storer N, Harrill D, Gerschenson M. Mitochondrial function, inflammation, fat and bone in HIV lipoatrophy: randomized study of uridine supplementation or switch to tenofovir. Antivir Ther. 2012;17(2):347-53. doi: 10.3851/IMP1928. Epub 2011 Oct 13. PMID 22293126
- See also: click here for more information about uridine supplementation or switch to tenofovir. — https://www.ncbi.nlm.nih.gov/pubmed/22293126/

RESULTS

PARTICIPANT FLOW:
Groups:
- Switch to TDF: Switch of AZT or d4T to tenofovir
  Tenofovir disoproxil fumarate: Switch thymidine NRTI to tenofovir
Period: Overall Study
Arm/Group | Uridine Supplementation | Switch to TDF
Started | 26 | 24
Completed | 22 | 23
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uridine Supplementation | Switch to TDF | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 48 [41 to 51] | 48 [43 to 51] | 48 [41 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 22 | 21 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat mtDNA Content
Description: Subcutaneous abdominal fat mitochondrial DNA (mtDNA)
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: copies/cell
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
copies/cell | -169 [-778 to 64] | 321 [-298 to 669]

2. Primary Outcome: Change in PBMC mtDNA
Description: Peripheral blood mononuclear cell (PBMC) mitochondrial DNA (mtDNA), measured in copies/cell
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: copies/cell
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
copies/cell | -24 [-158 to 91] | -52 [-105 to 108]

3. Secondary Outcome: Change in Limb Fat
Description: Change in limb fat as measured by dual-energy x-ray absorbtiometry (DEXA) scan
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: limb fat (kg)
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
limb fat (kg) | 0.1 [-0.03 to 0.3] | 0.4 [-0.06 to 1.2]

4. Secondary Outcome: Change in Trunk Fat
Description: Change in trunk fat as measured by dual-energy x-ray absorbtiometry (DEXA) scan
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: trunk fat (kg)
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
trunk fat (kg) | 0.2 [-0.5 to 0.6] | 0.7 [-0.04 to 1.4]

5. Secondary Outcome: Change in Lumbar Spine Bone Mineral Density (BMD)
Description: Change in lumbar spine bone mineral density (BMD) as measured by dual-energy x-ray absorbtiometry (DEXA) scan
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: lumbar spine BMD, g/cm^2
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
lumbar spine BMD, g/cm^2 | 0.39 [-0.96 to 1.68] | 0.0 [-2.9 to 1.76]

6. Secondary Outcome: Change in Hip Bone Mineral Density (BMD)
Description: Change in hip bone mineral density (BMD) as measured by dual-energy x-ray absorbtiometry (DEXA) scan
Time Frame: Baseline to Week 48
Measure: Median (Inter-Quartile Range); unit: hip BMD, g/cm^2
Arm/Group | Uridine Supplementation | Switch to TDF
Number analyzed (Participants) | 26 | 24
hip BMD, g/cm^2 | 0.45 [-0.27 to 3.56] | -3.3 [-5.1 to 0.0]

ADVERSE EVENTS:
Time Frame: Weeks 4,8,12,18 and 36
Description: Study evaluation was conducted at study entry and week 48; and additional safety visits were carried out at weeks 4,8,12,18 and 36 for the purpose of clinical and laboratory monitoring for toxicities, intolerance and adherance.
Arm/Group | Uridine Supplementation | Switch to TDF
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 8/26 | 6/24
Other Adverse Events (participants affected / at risk) | 18/26 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uridine Supplementation (N=26) | Switch to TDF (N=24)
Hypoglycemia Gr. 3 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abnormal phos. Gr. 3 (General disorders) | 1 (1) | 1 (3)
Renal calculus Gr. 3 (General disorders) | 1 (1) | 0 (0)
Elevated CK Gr. 3 & 4 (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Pancreatitis Gr. 3 (Endocrine disorders) | 0 (0) | 1 (1)
Vertigo Gr. 3 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypercholesterolem Gr. 3 (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea Gr. 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertrigliceridemia Gr. 3 & 4 (General disorders) | 2 (2) | 0 (0)
Abnormal AST Gr. 3 (General disorders) | 1 (1) | 0 (0)
Dysuria Gr. 3 (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uridine Supplementation (N=26) | Switch to TDF (N=24)
Incisional hematoma Gr. 1 & 2 (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Infected Incisional hematoma Gr. 2 (General disorders) | 0 (0) | 1 (1)
Incisional seroma Gr. 1 & 2 (General disorders) | 2 (2) | 1 (1)
Hyperglycemia Gr. 1 & 2 (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypoglycemia Gr. 1 & 2 (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophosphatemia Gr. 2 (General disorders) | 4 (6) | 4 (4)
Sinusitis Gr. 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia Gr. 2 (Cardiac disorders) | 0 (0) | 1 (1)
Thrombocytopenia Gr. 2 (Vascular disorders) | 1 (1) | 0 (0)
Elevated triglycerides Gr. 2 (General disorders) | 1 (1) | 1 (1)
URI Gr. 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated AST Gr. 2 (General disorders) | 1 (1) | 2 (2)
Diarhhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neurtropenia Gr. 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)
Otitis Gr. 2 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Prob. Herpes simplex Gr. 2 (General disorders) | 0 (0) | 1 (1)
Prob. Renal calculus Gr. 2 (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash/Bactrim allergy Gr. 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated CK Gr. 2 (General disorders) | 2 (3) | 1 (1)
Abnormal LDL Chol Gr. 2 (Vascular disorders) | 1 (1) | 0 (0)
Herpes zoster Gr. 2 (General disorders) | 0 (0) | 1 (1)
Incisional neuritis Gr. 2 (General disorders) | 1 (1) | 0 (0)
Gross hematuria Gr. 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal cholesterol Gr. 2 (Vascular disorders) | 1 (1) | 0 (0)
Abnormal Glucose Gr. 1 & 2 (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Abnormal ALT Gr. 2 (General disorders) | 0 (0) | 1 (1)
Abnormal BMD/T score Gr. 2 (General disorders) | 1 (1) | 0 (0)
Abnormal creatine Gr. 2 (General disorders) | 2 (2) | 0 (0)
Abnormal FBS Gr. 2 (General disorders) | 1 (1) | 0 (0)
Elevated LFTs Gr. 2 (General disorders) | 0 (0) | 1 (1)
Chalazion left eye - Gr. 2 (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size; Lack of control arm where tNRTI therapy was continued without any intervention; Adherence measured by sachet/pill count method.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No